CLINICAL TRIAL: NCT01001637
Title: Phase II Study of Curcumin Formulation (Longvida) or Placebo on Plasma Biomarkers and Mental State in Moderate to Severe Alzheimer's Disease or Normal Cognition
Brief Title: Efficacy and Safety of Curcumin Formulation in Alzheimer's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of support
Sponsor: Jaslok Hospital and Research Centre (Other)
Collaborators: Pharmanza Herbal Pvt Ltd (Unknown); Verdure Sciences (Industry); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dr Paresh Doshi, administrator, Jaslok Hospital and Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Longvida; 919820711140
Record Dates: First submitted 2009-10-15; First posted 2009-10-26 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Disease
Keywords: curcumin; alzheimer's; longVida; dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- curcumin (Active Comparator)
  Interventions: Dietary Supplement: Curcumin Formulation
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin Formulation — 2000mg or 3000mg daily BID
  Other Names: Longvida
  Arms: curcumin
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
Curcumin is shown to impact several different pathways of neuroprotection, however clinical trials have not shown positive results, due to the poor bioavailability of curcumin. This study is designed to determine efficacy and safety of high-bioavailability curcumin formulation (Longvida) in subjects with Alzheimer's disease.

DETAILED DESCRIPTION:
Curcumin is a polyphenolic molecule that comprises approximately 3-5% of turmeric (Curcuma longa) root, giving the spice its characteristic yellow color. Because of its anti-inflammatory, anti-amyloid, and antioxidant properties, curcumin has shown positive effects in animal models of Alzheimer's disease (AD). However, a six month human study was conducted with unformulated curcumin showing insignificant trends, due to limited bioavailability and brain permeability of unformulated curcumin. In animal models of AD, oral dosing of solid-lipid curcumin particle (SLCP or Longvida) significantly reduced memory deficit and impacted biomarkers better than unformulated curcumin. This study is to determine the potential efficacy and safety of highly absorbed SLCP curcumin in subjects with AD.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age ≥ 50.
* Diagnosed with probable AD using NINDS-ADRDA research criteria. MMSE score ≥5 and ≤20.
* No history of significant psychiatric or non-AD neurological disease.
* An available caregiver to monitor and administer medication and to accompany the subject to every clinical visit.
* On stable doses of concomitant medications for at least one month prior to starting study medication.

Exclusion Criteria:

* Current or recent major psychiatric illness that meets DSM-IV criteria (i.e. bipolar disorder, schizophrenia).
* Significant uncontrolled systemic illness (i.e. chronic renal failure, chronic liver disease, poorly controlled diabetes, or poorly controlled congestive heart failure).
* Recent history of gastrointestinal bleeding or ulceration.
* Alcoholism or substance abuse within the past year per DSM-IV criteria.
* Familial, autosomal dominant Alzheimer's disease due to a mutation in a known gene (Presenilin-1, Presenilin-2, or Amyloid Precursor Protein).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine if curcumin formulation affects mental capacity in Alzheimer's patients based on mental exams | 60 days

SECONDARY OUTCOMES:
To determine if curcumin formulation changes blood concentrations of amyloid-beta | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Fali Poncha, DM neuro, Study Director — Jaslok Hospital and Research Centre
Locations (1):
- Jaslok Hospital and research centre, Mumbai, Maharashtra, India